CLINICAL TRIAL: NCT00002965
Title: Phase II Study to Evaluate the Efficacy of Recombinant Interferon-Alpha in the Treatment of Recurrent Unresectable Meningiomas and Malignant Meningiomas
Brief Title: Interferon Alfa in Treating Patients With Recurrent Unresectable Meningiomas and Malignant Meningiomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM96-296; P30CA016672 (NIH); MDA-DM-96296 (Other: UT MD Anderson Cancer Center); NCI-G97-1206; CDR0000065463 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-07-11 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Interferon-alpha; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Benign Meningiomas (Experimental): INF alpha as a subcutaneous injection Monday to Friday for 8 weeks.
  Interventions: Biological: Recombinant Interferon Alfa (INF alpha)
- Arm 2: Other Pathologies (Experimental): INF alpha as subcutaneous injection Monday to Friday for 8 weeks.
  Interventions: Biological: Recombinant Interferon Alfa (INF alpha)

INTERVENTIONS:
Biological: Recombinant Interferon Alfa (INF alpha) — Subcutaneous injection Monday through Friday for 8 weeks.
  Other Names: Roferon; Interferon Alfa; Alpha 2 Interferon; IFN alpha-2A; IFN-Alpha 2; Interferon alfa 2a; Recombinant Interferon Alfa-2a

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells.

PURPOSE: Phase II trial to study the effectiveness of interferon alfa in treating patients with recurrent unresectable meningiomas and malignant meningiomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of recombinant interferon alpha (IFN alpha) as a single agent in the treatment of recurrent unresectable meningiomas and malignant meningiomas.
* Determine the nature and extent of central nervous system (CNS) toxicities associated with the use of alpha interferon in current doses and schedules.

OUTLINE: This is a two arm, randomized study. The first arm includes all histologically benign meningiomas. The second arm includes all other pathologies.

All patients receive INF alpha as a subcutaneous injection Monday through Friday for 8 weeks. Treatment continues without interruption as long as there is no tumor recurrence or progression and toxicity is acceptable.

Treatment continues without dose adjustment for the first 8 weeks as long as there are no toxic effects of grade III or greater. Dosage for subsequent courses is one dose level below the dose that produced toxicity of grade III or greater.

PROJECTED ACCRUAL: 20 patients will be entered per year into each arm.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven tumors:

  * Unresectable meningioma
  * Atypical meningioma
  * Malignant meningioma
  * Angioblastic meningioma
  * Hemangiopericytoma
* Recurrent or progressive, unresectable tumor after failing radiation therapy or refused radiation therapy following 2 surgeries

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Karnofsky at least 60%

Life expectancy:

* At least 3 months

Hematopoietic:

* AGC at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGPT less than 2.0 times normal
* Alkaline phosphatase less than 2.0 times normal
* Bilirubin less than 1.5 mg/dL

Renal:

* BUN less than 1.5 times normal OR
* Creatinine less than 1.5 times normal

Other:

* No active infection
* No diseases that obscure toxicity or dangerously alter drug metabolism
* No serious intercurrent medical illness
* Not pregnant
* Fertile patients must use adequate contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* Prior chemotherapy allowed and recovered from all myelotoxicity secondary to the therapy

Endocrine therapy:

* Prior hormonal therapy allowed
* No concurrent hormonal therapy

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1997-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity (DLT) | Each 8 weeks
  Efficacy of IFN alpha as single agent in treatment of recurrent unresectable/malignant meningiomas as measured by Dose Limiting Toxicities (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Kwan A. Yung, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org